CLINICAL TRIAL: NCT02474303
Title: A Demonstration Project of HIV Pre-exposure Prophylaxis (PrEP) With Tenofovir DF/Emtricitabine (TDF/FTC Among Female Sex Workers in Dakar, Senegal
Brief Title: Demonstration Project of PrEP Among Female Sex Workers in Dakar, Senegal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Réseau Africain de Recherche sur le SIDA (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Washington (Other); Westat (Other)
Responsible Party: Principal Investigator, Souleymane Mboup, Director, RARS, Réseau Africain de Recherche sur le SIDA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OPP1084414
Record Dates: First submitted 2015-04-03; First posted 2015-06-17 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: HIV/AIDS
Keywords: Truvada; EMTRICITABINE/TENOFOVIR DISPROXIL FUMARATE; HIV PREEXPOSURE PROPHYLAXIS (PrEP); Female Sex Workers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV Pre-exposure Prophylaxis (PrEP) (Other): Truvada
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Demonstration Study

SUMMARY:
Recent breakthroughs in antiretroviral (ARV)-based prevention provide new opportunities to rethink HIV prevention and treatment strategies, especially for key populations such as Female Sex Workers (FSWs). Antiretroviral (ARV)-based prevention of HIV transmission has the potential to have a profound population-level impact on the course of the HIV/AIDS pandemic. Several recently completed randomized controlled trials of HIV Pre-exposure Prophylaxis (PrEP) have shown efficacy at reducing HIV acquisition in high-risk populations. How to translate these trial results into population-level effects is the next critical step. PrEP "demonstration" projects, in collaboration with local stakeholders and at sites of routine care for high-risk populations provide an opportunity to move promising research results into actual public health benefits. With these key features in mind, the investigators propose an HIV PrEP demonstration project in FSW in Dakar, Senegal, West Africa. The objective of the proposed demonstration project with Tenofovir DF/Emtricitabine (TDF/FTC) among Female Sex Workers (FSW) in Dakar Senegal is to build a sustainable HIV PrEP program for FSW in Dakar, Senegal while demonstrating the feasibility of providing daily oral PrEP with Truvada (TDF/FTC) for 12 months to the enrolled FSW at Ministry of Heath run clinics (Pikine, Mbao, Rufisque and Diamniadio Health Centers). Critical milestones for this demonstration project with be feasibility, uptake, acceptability, use of TDF/FTC PrEP and programmatic retention of FSWs in Dakar MoH clinics. The investigators have assembled an expert team from RARS,The University of Washington, and Westat that have had greater than 2 decades of collaboration on HIV related projects in FSWs in Senegal. The investigators expect the results of this project will show that Senegal provides a unique opportunity to assess acceptability, feasibility, uptake and effectiveness of oral HIV PrEP at reducing HIV transmission in a high-risk FSW population.

DETAILED DESCRIPTION:
STUDY DESIGN This is a two-phase study, consisting of the following:

PHASE I - The feasibility evaluation for this study will take several forms.

* Observations - Field-based assessment of service delivery at each of the five sites;
* In-depth interviews - With policymakers, program managers, and service providers, as well as other community members and leaders; and
* Focus groups with registered and unregistered female sex workers (FSW). PHASE II - This will be a prospective demonstration study of oral pre-exposure prophylaxis (PrEP) with Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) for FSW with 12 months of follow up and a 3-month accrual period. A total of 267 FSW will be enrolled.

OBJECTIVES

Primary Objectives:

* Build a sustainable HIV PrEP program for FSW in Dakar, Senegal.
* Demonstrate the feasibility of providing daily oral PrEP with FTC/TDF for 12 months to FSW at Ministry of Health (MoH)-run clinics in Pikine, Mbao, Rufisque and Diamniadio Health Centers) in Dakar.

POPULATION & SAMPLE SIZE

PHASE I:

* 10 Key Informants: Policymakers, program managers, and service providers, as well as other community members and leaders.
* Focus Group Participants: 8 Registered and 8 Unregistered HIV-negative FSW age 18 or older.

PHASE II:

• 267 HIV-negative FSW age 18 or older recruited from four public health centers in Dakar: Pikine, Mbao, Rufisque and Diamniadio Health Centers.

PROTOCOL EVALUATIONS

* PHASE I: Qualitative data from observations, key informant interviews, and focus groups will be collected, analyzed and used to inform the implementation of Phase II.
* PHASE II: Quantitative data will be collected using behavioral measures and clinical and laboratory evaluations. Data from electronic monitoring will also be collected.

STUDY DURATION 24 months

REGIMEN Daily oral PrEP with FTC/TDF for 12 months

ELIGIBILITY:
Inclusion Criteria:

* • Completion of the written informed consent process prior to undergoing any screening evaluations

  * ≥ 18 years and older
  * Active sex work (Paid sex within the past six months)
  * In general good health, confirmed by medical history and physical examination
  * Has laboratory evidence of absence of HIV infection, defined as a negative 4th generation HIV ELISA test prior to enrollment
  * Serum creatinine less than or equal to the upper limit of normal (ULN) and calculated creatinine clearance of at least 70 mL/minute by Cockcroft-Gault formula
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 2.5 times ULN
  * Hemoglobin greater than 8.5 g/dL
  * Does not report intention to relocate out of the study area during the course of the study
  * If able to become pregnant, self-reported use of an effective method of contraception at enrollment, and intending to use an effective method during the follow-up period
  * Without signs or symptoms of acute HIV infection (acute retroviral syndrome)

Exclusion Criteria:

* • HIV-1 and HIV-2 screening tests are reactive

  * Is enrolled in any other clinical product trial
  * Serious and active medical condition
  * Proteinuria 2+ or greater at screening
  * Glucosuria 2+ or greater at screening
  * Use of disallowed medications (*See note below)
  * Presence of active serious psychiatric symptoms (e.g., active hallucinations, suicidal, homicidal, or exhibiting violent behavior) at the time of consent
  * Intoxicated or under the influence of alcohol or other drugs at the time of screening
  * Pregnant females and females who are breast-feeding
  * Any other reason or condition that in the opinion of the investigator would interfere with participation, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The number/proportion of FSWs who remain in the program | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Souleymane Mboup, Ph.D., Principal Investigator — RARS; Geoffrey S Gottlieb, M.D, Principal Investigator — University of Washington; Moussa Sarr, M.D., MPH, Principal Investigator — Westat
Locations (4):
- Senegal (4):
  - Centre de santé de Mbao, Dakar
  - Centre de Santé de Rufisque, Dakar
  - Centre de Santé Dominique de Pikine, Dakar
  - centre hospitalier de Diamniadio, Dakar